CLINICAL TRIAL: NCT04956939
Title: Levodopa Response and Gut Microbiome in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Director of Center for Integrated Microbiome and Chronobiology Research, Rush University Medical Center
Other Study IDs: RUMC 18032006
Record Dates: First submitted 2021-06-11; First posted 2021-07-09 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: levodopa
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool collection, saliva and oral swab, breath test, blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: PD patients receiving low frequency dose of levodopa.
  Interventions: Drug: Low dose levodopa
- Group 2: PD patients receiving high frequency dose of levodopa.
  Interventions: Drug: High dose levodopa
- Control Group: Spouses of PD patients without PD diagnosis

INTERVENTIONS:
Drug: Low dose levodopa — Low frequency is defined as ≤ 3 LD doses a day
  Groups: Group 1
Drug: High dose levodopa — High frequency dosage is defined as ≥ 5 LD doses per day
  Groups: Group 2

SUMMARY:
Levodopa (LD) is an effective treatment to control symptoms of Parkinson's disease (PD). However, the response to (the effectiveness) LD changes over time and patients require higher and more frequent LD doses for treatment. The purpose of this study is to identify what reasons or causes might influence the changes in LD effectiveness, particularly if intestinal bacteria contribute to the breakdown of LD in patients with PD. This study is an observational cohort proof-of-concept study that follows PD patients who take PD at high-frequency doses and low-frequency doses. . Each PD patient will have a household healthy control/spouse enrolled into the study. Single patients with no spouse will still be eligible to enroll.

DETAILED DESCRIPTION:
Levodopa (LD) is an effective treatment to control symptoms of Parkinson's disease (PD) and during the first few years of LD treatment patients are said to experience a 'honeymoon' period, reflective of a sustained beneficial response to this dopamine pro-drug. However, the response to LD changes over time and patients require higher and more frequent LD doses. Most patients develop motor response complications such as frequent periods of immobility and involuntary movements. The major unmet need is to preserve the initial, stable, response to LD and prevent the development of motor response complications. It is therefore essential to identify the underlying mechanism for the changes in LD effectiveness.

This study involves only 1 study visit. Prior to the study visit, participants will be asked to complete questionnaires and will receive an at-home stool collection kit. At the time of the study visit, participants will turn in their questionnaires and their at-home stool sample. On the day of the study visit, the patient will have fasted (overnight for 8 hours) and taken their last LD medication 12 hours prior to the visit. Each patient (and healthy control) will bring a home collected stool sample to their scheduled research visit which will be taken and stored in -80 freezers for the microbiota analysis. Oral swab will be collected for oral microbiota analysis. For PD patients only, an indwelling catheter for blood draws will be placed by one of the highly experienced GI infusion nurses and a fasting blood sample will be drawn. At the time of the visit, each patient will be given their morning LD dose (1.5 times their usual dose as they did not take LD for 12 hours), and then both patients and their controls will be given lactulose (20 mg) and have their breath collected every 10 minutes for the first hour, and then every 15 minutes for the following 3 hours (total 4 hours) for measurement of breath hydrogen and methane to assess mouth to cecum transit and presence/absence of small bowel bacteria overgrowth. PD patients will also have a blood sample drawn every 30 minutes, for 4 hours (total 8 draws) to measure LD and LD metabolites in the plasma Patients and controls will be provided a light breakfast (2 white wheat bread toasts with thin layer of butter and coffee). Each patient and control will complete a detailed dietary questionnaire (FFQ and 24 hour diet recall), a food timing questionnaire and screener and a structured demographic questionnaire. PD patients will also complete a questionnaire that includes PD-related information. Patients will also perform a simple finger tapping task to asses and quantify speed of movement before, during and after completion of study. Finger tapping task will be done using 2 mechanical counters mounted on a board. The patients go back and forth between these two counters and the number of taps in 30 seconds will be automatically recorded. In addition, patients will log their motor state (OFF versus ON) every half an hour on a PD diary.

ELIGIBILITY:
FOR PATIENTS WITH PD:

Inclusion Criteria:

* Documented diagnosis of Parkinson's disease
* On Levodopa treatment

Exclusion Criteria:

* History of GI diseases [except for hemorrhoids or occasional (<3 times a week) heartburn] like Inflammatory bowel disease or Celiac disease
* Antibiotic use within last 12 weeks
* Use of probiotic supplement over the prior 2 weeks except yogurt
* Intentional change in diet
* Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study. Low does aspirin is allowed.

FOR CONTROL GROUP:

Inclusion Criteria:

* No clinical evidence of neurological disorders including Parkinson's disease
* Live in the same household as the Parkinson's Disease patient or is a first degree relative of the PD patient.

Exclusion Criteria:

* History of GI diseases [except for hemorrhoids or occasional (<3 times a week) heartburn] like Inflammatory bowel disease or Celiac disease
* Antibiotic use within last 12 weeks
* Use of probiotic supplement over the prior 2 weeks except yogurt
* Intentional change in diet
* Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study. Low does aspirin is allowed.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to enroll two groups of established PD patients on a stable dose of LD for the prior 4 weeks. We will enroll twelve patients in each of the following two groups: Group 1:"low frequency dose" patients and Group 2:" high frequency dose "patients. Low frequency is defined as ≤ 3 LD doses a day and high frequency as ≥ 5 LD doses per day. Each PD patient will have a household healthy control/spouse enrolled into the study. Single patients with no spouse will still be eligible to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Fecal microbial community structure and functional changes for phylum, genus and species taxonomic level bacteria, virus, fungi, and archaea. | During the study visit,1 day
  Quantitative polymerase chain reaction (qPCR), 16S rRNA Sequencing and Shotgun Metagenomics
Oral microbial community structure and functional changes for phylum, genus and species taxonomic level bacteria, virus, fungi, and archaea. | During the study visit,1 day
  Quantitative polymerase chain reaction (qPCR), 16S rRNA Sequencing and Shotgun Metagenomics
Change in the measurement of blood biomarker levodopa (ng/mL) over 12 time frames | During the study visit,1 day
  ELISA (enzyme-linked immunosorbent assay)
Change in the measurement of blood biomarker glucagon-like peptide-1 (GLP-1) (pm) over 12 time frames | During the study visit,1 day
  ELISA (enzyme-linked immunosorbent assay)
Change in the measurment scores of breath hydrogen and methane to assess mouth to cecum transit and presence or absence of small bowel bacteria overgrowth over 16 time frames. | During the study visit,1 day
  Lactulose Breath Scoring Test
Change in the measurement of blood levodopa metabolomics concentrations (ug/mL) across 12 time frames. | During the study visit,1 day
  Gas Chromatography - Tandem Mass Spectrometry (GC-MS/MS)
Changes in the measurement of blood targeted short chain fatty acids (SCFA) metabolomics concentrations (ug/mL) for acetate, propionate, butyrate and total SCFA across 12-time frames | During the study visit,1 day
  Gas Chromatography - Tandem Mass Spectrometry (GC-MS/MS)
Change in the measurement of blood targeted trimethylamine N-oxide (TMAO) concentrations (uM) across 12 time frames | During the study visit,1 day
  Liquid Chromatography-Mass Spectrometry (LC-MS/MS)

SECONDARY OUTCOMES:
Food Timing Screener | During the study visit,1 day
  Food Timing Screener (FTS) questionnaire. A structured food demographics questionnaire was therefore developed to access food timing. The questionnaire consists of eight questions asking subjects' eating habits on work days and non-work days. Questions include the time of the main meal during work and non-work days, time of last meal before bed, consistency of dinner within work and non-work days, and consistency of breakfast, lunch, and dinner between work and non-work days.
Food and Frequency of Consumption | During the study visit,1 day
  Food Timing Questionnaires (FTQ) consists of a list of foods and the frequency in which these foods are consumed.
Single day food recall | During the study visit,1 day
  Automated Self-Administered 24-Hour Recall (ASA24) Dietary Assessment. Total nutrients from all supplements reported in a given day.
Gastrointestinal Symptom and Severity | During the study visit,1 day
  Patient-Reported Outcomes Measurements Information System (PROMIS) gastrointestinal questionnaire for Belly Pain (6 questions), Bowel Incontinence (4 questions), Constipation (9 questions), and Gas & Bloating (12 questions). Higher score denoted more GI symptoms. Lower score denotes less GI symptoms. Scores range from 20 (low) to 80 (high). A score of 50 is denoted as the general population.
Diet change | During the study visit,1 day
  Vioscreen Food Frequency Questionnaire (FFQ). Total of 19 measured food components. Vioscreen captures comprehensive dietary behaviors in just 30 minutes. It is a unique dietary questionnaire, management and analysis system that efficiently gathers and manages data that immediately identifies dietary "habits" and counsel for lifestyle changes.
REM Sleep Behavior Disorder assessment | During the study visit,1 day
  RBD1Q questionnaire that consists of a single question, answered "yes" or "no," as follows: "Have you ever been told, or suspected yourself, that you seem to 'act out your dreams' while asleep (for example, punching, flailing your arms in the air, making running movements, etc.)?"
Sleep Disturbance | During the study visit,1 day
  The Patient Reported Outcomes Measurement Information System (PROMIS) is a self-reported questionnaire that assess the sleep-wake function in adults.
Chronotype | During the study visit,1 day
  The Munich ChronoType Questionnaire (MCTQ) uses a self-rated scale to assess individual phase of entrainment on work and work-free days; it is a tool to collect primary sleep times, such as bed- and rise-times, plus the clock time of becoming fully awake as well as sleep latency and inertia, in addition to other time points.
Functional status in patients with Parkinson's Disease | During the study visit,1 day
  The On-Off Parkinson's Disease Diary by Hauser assesses troublesome and non-troublesome dyskinesia through self-reported time markers.
Motor speed and lateralized coordination | During the study visit,1 day
  PD patients will take a Finger-Tapping Test (FTT) where hands are laid flat and fingers are lifted one at a time onto two mechanical counters mounted on a board. The patients go back and forth between these two counters and the number of taps in 30 seconds will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States